CLINICAL TRIAL: NCT02044874
Title: A 12-Week, Multicenter, Double-blind, Randomized, Placebo-controlled Parallel-group Phase 2 Dose Selection Study of Lorcaserin Hydrochloride, an Oral 5-HT2C Receptor Agonist for Smoking Cessation
Brief Title: A Study to Evaluate the Effect of Lorcaserin Hydrochloride on Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-035
Record Dates: First submitted 2014-01-21; First posted 2014-01-24 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- APD356 10 mg b.i.d. (Experimental): APD356 - lorcaserin hydrochloride 10 mg tablet administered twice daily for 12 weeks
  Interventions: Drug: APD356-lorcaserin hydrochloride
- APD356 10 mg q.d. (Experimental): APD356 - lorcaserin hydrochloride 10 mg tablet administered once daily and one matching placebo tablet administered once daily for 12 weeks
  Interventions: Drug: APD356-lorcaserin hydrochloride
- Placebo 10 mg b.i.d (Placebo Comparator): Placebo tablet matching the APD356-lorcaserin hydrochloride 10 mg tablet administered twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD356-lorcaserin hydrochloride
  Other Names: Belviq
  Arms: APD356 10 mg b.i.d.; APD356 10 mg q.d.
Drug: Placebo
  Arms: Placebo 10 mg b.i.d

SUMMARY:
In smokers who are motivated to stop smoking, treatment with lorcaserin compared with placebo will provide greater abstinence as measured by the last 4 weeks of treatment (Weeks 9-12). The target quit date was Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-65 years, inclusive
2. ≥10 cigarettes per day with no period of abstinence longer than 3 months in the past year and who are motivated to quit smoking
3. Able to give signed informed consent
4. Eligible female patients will be:

   1. non-pregnant
   2. non-lactating
   3. agree to use an acceptable method of effective contraception during the study
5. Eligible male patients agree to use contraception when sexually active with a female partner who is not using an acceptable method of birth control
6. Body weight of ≥50 kg (110 pounds), inclusive
7. Considered to be in stable health in the opinion of the investigator

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Prior or current use of lorcaserin HCl
2. Prior participation in any study of a nicotine vaccination
3. Use of other therapies for smoking cessation is not allowed within 3 months of screening through study exit
4. Use of tobacco products other than cigarettes
5. Prior use of fenfluramine or dexfenfluramine
6. Serious or unstable medical condition or clinically significant new illness within the 6 months prior to screening
7. Previous participation in any clinical study within 6 weeks prior to the screening visit
8. History of severe allergies, severe drug or excipient allergy or hypersensitivity
9. History of significant cardiovascular condition
10. History of other significant medical conditions
11. Significant risk of suicide
12. Anticipated use of any agents that are associated with valvulopathy and/or pulmonary hypertension
13. Positive test result for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
14. Recent history of alcohol or drug/solvent abuse
15. Concurrent participation in the study by more than one member of the same household
16. Not suitable to participate in the study in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Anderson, M.D., Principal Investigator — Desert Valley Research; Rancho Mirage, California
Locations (31):
- United States (31):
  - Pharmacology Research Institute, Encino, California
  - Synergy Escondido, Escondido, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Desert Valley Research, Rancho Mirage, California
  - Avail Clinical Research, DeLand, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Compass Research East, Leesburg, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, Orlando, Florida
  - Compass Research East, Oviedo, Florida
  - Meridien Research, Tampa, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Integrative Clinical Trials, Brooklyn, New York
  - Duke University, Durham, North Carolina
  - PMG Research Inc., Raleigh, North Carolina
  - PMG Research Inc., Wilmington, North Carolina
  - PMG Research Inc., Winston-Salem, North Carolina
  - Neurobehavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Clinical Trial Center, Jenkintown, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - KRK Medical Research, Dallas, Texas

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Shanahan WR, Rose JE, Glicklich A, Stubbe S, Sanchez-Kam M. Lorcaserin for Smoking Cessation and Associated Weight Gain: A Randomized 12-Week Clinical Trial. Nicotine Tob Res. 2017 Aug 1;19(8):944-951. doi: 10.1093/ntr/ntw301. PMID 27815511

RESULTS

PARTICIPANT FLOW:
Groups:
- APD356 10 mg b.i.d.; APD356 10 mg q.d.: APD356-lorcaserin hydrochloride
- Placebo 10 mg b.i.d: Placebo
Period: Overall Study
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo 10 mg b.i.d
Started | 201 | 202 | 200
Completed | 171 | 147 | 140
Not Completed | 30 | 55 | 60
Not completed — Adverse Event | 5 | 6 | 6
Not completed — Withdrawal by Subject | 8 | 16 | 23
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Lost to Follow-up | 10 | 27 | 21
Not completed — Sponsor Decision | 0 | 1 | 1
Not completed — Other | 7 | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- APD356 10 mg b.i.d.: APD356-lorcaserin hydrochloride 10 mg twice daily
- APD356 10 mg q.d.: APD356-lorcaserin hydrochloride 10 mg once daily
- Placebo 10 mg b.i.d: Placebo 10 mg twice daily
- Total: Total of all reporting groups
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo 10 mg b.i.d | Total
Number analyzed (Participants) | 201 | 202 | 200 | 603
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 200 | 200 | 198 | 598
  >=65 years | 1 | 2 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.3) | 45.0 (11.3) | 46.3 (11.7) | 45.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 100 | 118 | 328
  Male | 91 | 102 | 82 | 275
Region of Enrollment [Number; unit: participants]
  United States | 201 | 202 | 200 | 603

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Abstinence for the Last 4 Weeks of Treatment From Weeks 9-12
Description: Primary efficacy was assessed as the CO (carbon monoxide)-confirmed continuous abstinence rate for the last 4 weeks of treatment (Month 3: Weeks 9 through 12), defined as no reported smoking (not even a puff) or other nicotine use, verified by end expiratory CO levels <= 10 ppm.
Time Frame: Week 9 - Week 12
Population: Modified Intent-to-Treat: All randomized patients, who received at least 1 dose of study medication, had a baseline measurement, and have a post-randomization measurement
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Number analyzed (Participants) | 196 | 195 | 195
percentage of participants | 15.31 | 8.72 | 5.64
Statistical Analysis 1: Comparison: APD356 10 mg b.i.d. vs Placebo; Test type: Superiority or Other; p = 0.0027, Regression, Logistic; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.47 to 6.22]
Statistical Analysis 2: Comparison: APD356 10 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.2427, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.73 to 3.51]
Statistical Analysis 3: Comparison: APD356 10 mg b.i.d. vs APD356 10 mg q.d; Test type: Superiority or Other; p = 0.0477, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.01 to 3.56]

2. Secondary Outcome: Abstinence During Weeks 3-12
Description: The CO (carbon monoxide)-confirmed continuous abstinence rate for Weeks 3 through 12, defined as no reported smoking (not even a puff) or other nicotine use, verified by end expiratory CO levels <= 10 ppm
Time Frame: Week 3 to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Number analyzed (Participants) | 196 | 195 | 195
percentage of participants | 5.61 | 3.59 | 2.05
Statistical Analysis 1: Comparison: APD356 10 mg b.i.d. vs Placebo; Test type: Superiority or Other; p = 0.0784, Regression, Logistic; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.89 to 9.08]
Statistical Analysis 2: Comparison: APD356 10 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.3650, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.51 to 6.17]
Statistical Analysis 3: Comparison: APD356 10 mg b.i.d. vs APD356 10 mg q.d; Test type: Superiority or Other; p = 0.3438, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.61 to 4.21]

3. Secondary Outcome: The 7 Day Point Prevalence or Weekly Abstinence at Week 8
Description: The CO (carbon monoxide)-confirmed continuous abstinence rate at for the 7-day period preceding the Week 8 visit, defined as no reported smoking (not even a puff) or other nicotine use, verified by end expiratory CO levels <= 10 ppm
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Number analyzed (Participants) | 196 | 195 | 195
percentage of participants | 16.33 | 9.74 | 9.23
Statistical Analysis 1: Comparison: APD356 10 mg b.i.d. vs Placebo; Test type: Superiority or Other; p = 0.0379, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.04 to 3.55]
Statistical Analysis 2: Comparison: APD356 10 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.8628, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.54 to 2.09]
Statistical Analysis 3: Comparison: APD356 10 mg b.i.d. vs APD356 10 mg q.d; Test type: Superiority or Other; p = 0.0556, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.99 to 3.31]

4. Secondary Outcome: The 7 Day Point Prevalence or Weekly Abstinence at Week 12
Description: The CO (carbon monoxide)-confirmed continuous abstinence rate at for the 7-day period preceding the Week 12 visit, defined as no reported smoking (not even a puff) or other nicotine use, verified by end expiratory CO levels <= 10 ppm
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of paticipants
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Number analyzed (Participants) | 196 | 195 | 195
percentage of paticipants | 20.41 | 13.85 | 11.79
Statistical Analysis 1: Comparison: APD356 10 mg b.i.d. vs Placebo; Test type: Superiority or Other; p = 0.0219, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.10 to 3.35]
Statistical Analysis 2: Comparison: APD356 10 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.5450, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.66 to 2.18]
Statistical Analysis 3: Comparison: APD356 10 mg b.i.d. vs APD356 10 mg q.d; Test type: Superiority or Other; p = 0.0868, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.93 to 2.72]

5. Secondary Outcome: Body Weight
Description: Change in body weight from Week 1 (baseline) to Week 12
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Kg
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Number analyzed (Participants) | 170 | 150 | 141
Kg | -0.98 [-1.35 to -0.61] | -0.35 [-0.74 to 0.04] | -0.01 [-0.40 to 0.38]
Statistical Analysis 1: Comparison: APD356 10 mg b.i.d. vs Placebo; Test type: Superiority or Other; p = 0.0004, Mixed-effects repeated measures; Difference in LS Means = -0.97, 95% CI 2-sided [-1.51 to -0.43]
Statistical Analysis 2: Comparison: APD356 10 mg q.d. vs Placebo; Test type: Superiority or Other; p = 0.2268, mixed effects repeated measures; Difference in LS Means = -0.34, 95% CI 2-sided [-0.89 to 0.21]
Statistical Analysis 3: Comparison: APD356 10 mg b.i.d. vs APD356 10 mg q.d; Test type: Superiority or Other; p = 0.0217, mixed effects repeated measures; Difference in LS Means = -0.63, 95% CI 2-sided [-1.17 to -0.09]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening through the follow-up visit at Week 14 for a total period of up to 17 weeks.
Arm/Group | APD356 10 mg b.i.d. | APD356 10 mg q.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 3/201 | 4/202 | 1/200
Other Adverse Events (participants affected / at risk) | 70/201 | 65/202 | 68/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD356 10 mg b.i.d. (N=201) | APD356 10 mg q.d. (N=202) | Placebo (N=200)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood carbon monoxide increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD356 10 mg b.i.d. (N=201) | APD356 10 mg q.d. (N=202) | Placebo (N=200)
Nausea (Gastrointestinal disorders) | 16 (16) | 9 (9) | 10 (10)
Constipation (Gastrointestinal disorders) | 12 (12) | 13 (13) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 7 (7) | 6 (6)
Fatigue (General disorders) | 11 (11) | 6 (6) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 8 (8) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 6 (6) | 8 (8)
Headache (Nervous system disorders) | 19 (19) | 23 (23) | 16 (16)
Dizziness (Nervous system disorders) | 9 (9) | 11 (11) | 4 (4)
Abnormal dreams (Psychiatric disorders) | 8 (8) | 8 (8) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 5 (5) | 8 (8)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3) | 5 (5)
Irritability (Psychiatric disorders) | 2 (2) | 3 (3) | 8 (8)

LIMITATIONS AND CAVEATS:
Demonstration of sustained abstinence requires a study of >12 weeks duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less